CLINICAL TRIAL: NCT03637387
Title: A Phase 3 Placebo-Controlled, Double-Blind Randomized Withdrawal Study to Evaluate the Efficacy and Safety of BIIB074 in Subjects With Trigeminal Neuralgia
Brief Title: 802NP302 Efficacy and Safety Study of BIIB074 in Participants With Trigeminal Neuralgia
Acronym: SURGE-2
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 802NP302; 2016-002473-35 (EudraCT Number)
Record Dates: First submitted 2018-08-16; First posted 2018-08-20 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Trigeminal Neuralgia
Keywords: TGN; TN
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — vixotrigine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- BIIB074 (Experimental): Administered orally three times daily (TID)
  Interventions: Drug: BIIB074
- Placebo (Placebo Comparator): Placebo matching BIIB074
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIB074 — Administered as specified in the treatment arm
  Arms: BIIB074
Drug: Placebo — Administered as specified in the treatment arm.
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the efficacy of BIIB074 in treating pain experienced by participants with trigeminal neuralgia (TN).

The secondary objectives are to investigate the safety and tolerability of BIIB074 in participants with TN and to evaluate the population pharmacokinetic(s) (PK) of BIIB074.

ELIGIBILITY:
Key Inclusion Criteria:

* A diagnosis of trigeminal neuralgia (TN) for at least 3 months based on International Headache Society (IHS) diagnostic criteria.
* Participant must have failed at least 1 prior standard of care pharmacologic treatment for TN (defined as an inadequate response or intolerance to treatment), as determined by the Investigator based on medical history.
* Age ≥18 years at the time of informed consent.
* Participants must have recorded their pain score in their eDiary on at least 5 days during the run-in period (Days -7 to -1).
* Allowed concomitant medications must have been stable for at least 4 weeks prior to Day 1 of the dose-optimization period. The maximum dosage of carbamazepine allowed on Day 1 is 400 mg/day (or 600 mg/day for oxcarbazepine).

Key Exclusion Criteria:

* History or positive test result at Screening for hepatitis C virus antibody or current hepatitis B infection (defined as positive for hepatitis B surface antigen [HBsAg] and/or hepatitis B core antibody [HBcAb]).
* Positive history of human immunodeficiency virus (HIV) or a positive HIV test at Screening.
* Participants with facial pain other than TN.
* Personal or family (first-degree relative) history of seizures (except for simple febrile convulsions) or clinically significant head injury.
* Positive drug screen for drugs of abuse at Screening (amphetamine [methamphetamines and 3,4-methylenedioxymethamphetamine], phencyclidine, barbiturates, benzodiazepines, cocaine, opioids) except if explained by use of allowed prescription medicines. Prospective subjects with a positive screen for tetrahydrocannabinol must agree to discontinue use upon study enrollment and for the duration of the study.
* Known hypersensitivity to BIIB074 or components of the BIIB074 formulation or matching placebo.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2025-08-18 (Estimated); Study Completion 2026-09-29 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Classified as Responders at Week 12 of the Double- Blind Period | Week 12
  A participant who meets all of the following criteria will be classified as a responder: (1) Has a reduction of >=30% in mean pain score compared with baseline; (2) Has not discontinued randomized treatment before the end of Week 12 of the double-blind period; (3) Has not taken prohibited pain medication before the end of Week 12 of the double-blind period.
Number of Participants Experiencing Adverse Events (AEs) and Serious Adverse Events (SAEs) During the Long Term Extension (LTE) Period | Baseline up to Week 52 of the LTE
  An AE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. An SAE was defined as any untoward medical occurrence that at any dose: results in death; in the view of the Investigator, places the subject at immediate risk of death (a life-threatening event; however, this does not include an event that, had it occurred in a more severe form, might have caused death); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; or results in a congenital anomaly/birth defect.

SECONDARY OUTCOMES:
Percentage of Participants Classified as Responders Achieving Patient Global Impression of Change (PGIC) Response at Week 12 of the Double-Blind Period | Week 12
  A participant who meets all of the following criteria will be classified as a responder: (1) Achieving Patient Global Impression of Change (PGIC) response of "Much Improved" or "Very Much Improved" at Week 12 of the double-blind period; (2) has not discontinued randomized study treatment before the end of Week 12 of the double-blind period; (3) has not taken prohibited pain medication before the end of Week 12 of the double-blind period. PGIC is a 7-item self-report scale depicting a participant's rating of overall improvement. Participants rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."
Percentage of Participants Classified as Responders Achieving >=50 Percent Reduction From Baseline Mean Number of Paroxysms at Week 12 | Week 12
  A participant who meets all of the following criteria will be classified as a responder: (1) Achieving >=50 percent reduction from baseline mean number of paroxysms at Week 12; (2) has not discontinued randomized study treatment before the end of Week 12 of the double-blind period; (3) has not taken prohibited pain medication before the end of Week 12 of the double-blind period. A paroxysm is a trigeminal neuralgia pain attack.
Percentage of Participants Classified as Responders Achieving >=50 Percent Reduction From Baseline Mean Pain Score at Week 12 | Week 12
  A participant who meets all of the following criteria will be classified as a responder: (1) Achieving >=50 percent reduction from baseline mean pain score at Week 12; (2) has not discontinued randomized study treatment before the end of Week 12 of the double-blind period; (3) has not taken prohibited pain medication before the end of Week 12 of the double-blind period. Pain score is a 11-point numerical rating scale where 0 = no pain; 10 = maximum pain imaginable. Higher scores representing more pain.
Number of Participants Experiencing Adverse Events (AEs) and Serious Adverse Events (SAEs) During the Double Blind Period | Up to Week 14 of Double blind period
  An AE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. An SAE was defined as any untoward medical occurrence that at any dose: results in death; in the view of the Investigator, places the subject at immediate risk of death (a life-threatening event; however, this does not include an event that, had it occurred in a more severe form, might have caused death); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; or results in a congenital anomaly/birth defect.
Area Under the Plasma Concentration- Time Curve at Steady State (AUC,ss) | Day 15, 29, 43, 57, 71, 85, 99, 113, 127, 141, premature treatment discontinuation (if occurred)
  AUC,ss= Area under the plasma concentration versus time curve (AUC) at steady state.
Maximum Observed Plasma Concentration at Steady State (Cmax,ss) | Day 15, 29, 43, 57, 71, 85, 99, 113, 127, 141, premature treatment discontinuation (if occurred)
  Cmax,ss= Maximum Observed Plasma Concentration of BIIB074 at Steady State
Percentage of Participants with >=30% Reduction From Baseline in Mean Pain Score During the Long Term Extension (LTE) Period | Week 1 through Week 52
  Pain score is a 11-point numerical rating scale where 0 = no pain; 10 = maximum pain imaginable. Higher scores representing more pain.
Change From Baseline in Mean Pain Score During the Long Term Extension (LTE) Period | Baseline, Week 1 through Week 52
  Pain score is a 11-point numerical rating scale where 0 = no pain; 10 = maximum pain imaginable. Higher scores representing more pain.
Change From Baseline in Mean Worst Pain Score During the Long Term Extension (LTE) Period | Baseline, Week 1 through Week 52
  Pain score is a 11-point numerical rating scale where 0 = no pain; 10 = maximum pain imaginable. Higher scores representing more pain.
Percentage of Participants with >=50% Reduction From Baseline in Mean Number of Paroxysms During Long Term Extension (LTE) Period | Week 1 through Week 52
  Paroxysms are trigeminal neuralgia pain attacks. They are short, severe, and sharp, shooting, stabbing, or shock-like.
Change From Baseline in Mean Number of Paroxysms During Long Term Extension (LTE) Period | Baseline, Week 1 through Week 52
  Paroxysms are trigeminal neuralgia pain attacks. They are short, severe, and sharp, shooting, stabbing, or shock-like.
Percentage of Participants With a PGIC Response of "Much Improved or "Very Much Improved" by Visit During the Long Term Extension (LTE) Period | Day 1, Week 2, 4, 6, 8, every 12 weeks up to Week 52
  PGIC is a 7-point self-report scale depicting a participant's rating of overall improvement. Participants rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse." Participants with "Much Improved or "Very Much Improved" will be reported.
Change From Baseline in the PENN-FPS-R Score by Visit During the Long Term Extension (LTE) Period | Baseline, Day 1, Week 2, 4, 6, 8, every 12 weeks up to Week 52
  The Penn-FPS-R is a new 12-item Health-Related Quality of Life outcome measure with content validity that can be used to assess and monitor the impact of Trigeminal Neuralgia and facial pain treatment interventions in both clinical practice and research. This scale uses the 0-10 numeric rating scale (NRS) to quantify the pain impact different activities and quality of life items, where 0 indicates no interference and 10 indicates complete interference. The sum of the rated NRS score will be calculated.
Change From Baseline in the EQ-5D-5L Score by Visit During the Long Term Extension (LTE) Period | Baseline, Day 1, Week 4, 8, every 12 weeks up to Week 52
  EQ-5D-5L is a standardized, subject-rated instrument for use as a measure of health outcomes. The EQ 5D-5L includes 2 components: the EQ-5D-5L descriptive system and the EQ-Visual Analog Scale (EQ-VAS). The EQ-5D-5L descriptive system provides a profile of the participant's health state in 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). For each dimension, the participant is instructed to indicate whether he or she has no problems, slight problems, moderate problems, severe problems, and extreme problems. A negative change from Baseline indicates improvement.
Change From Baseline in the WPAI Neuropathic Pain (V2.0) Score by Visit During the Long Term Extension (LTE) Period | Baseline, Day 1, Week 4, 8, every 12 weeks up to Week 52
  The WPAI questionnaire is a validated instrument to measure impairments in work and activities. The WPAI yields four types of scores: 1. Absenteeism (percentage of work time missed) 2. Presenteeism (percentage of impairment at work/reduced on-the-job effectiveness) 3. Work productivity loss (percentage of overall work impairment [absenteeism plus presenteeism]) 4. Activity Impairment (percentage of overall activity impairment). WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/